CLINICAL TRIAL: NCT05440435
Title: Application of Mobile DR in the Diagnosis of Bone Trauma in High Cold Environment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rongrong Hua (Other)
Responsible Party: Sponsor-Investigator, Rongrong Hua, Principal Investigator, General Hospital of Chinese Armed Police Forces
Organization: General Hospital of Chinese Armed Police Forces (Other)
Other Study IDs: DR001
Record Dates: First submitted 2022-06-24; First posted 2022-06-30 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Bone Injury; Artificial Intelligence
Keywords: Artificial intelligence; Digital radiography
MeSH Terms: interventions — Radiographic Image Enhancement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Center A: Study center A that observe cohort populations (sample size=400).
  Interventions: Diagnostic Test: digital radiography (DR)
- Center B: Study center B that observe cohort populations (sample size=400).
  Interventions: Diagnostic Test: digital radiography (DR)
- Center C: Study center C that observe cohort populations (sample size=400).
  Interventions: Diagnostic Test: digital radiography (DR)
- Center D: Study center D that observe cohort populations (sample size=400).
  Interventions: Diagnostic Test: digital radiography (DR)
- Center E: Study center E that observe cohort populations (sample size=400).
  Interventions: Diagnostic Test: digital radiography (DR)

INTERVENTIONS:
Diagnostic Test: digital radiography (DR) — Patients with bone injury received routine and mobile DR sequential examination.

SUMMARY:
In the high cold environment, mobile digital radiography (DR) is used to collect the imaging of bone injury patients, and the artificial intelligence diagnosis module is used to diagnose the injury. The quality of images obtained by mobile or conventional DR and the consistency between artificial intelligence and pure artificial diagnosis will be analyzed respectively. Finally, the application value of mobile DR loaded with artificial intelligence diagnosis function in high cold environment is determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients with new bone injury

Exclusion Criteria:

* Life threatening.
* Head injury and fracture.
* There are congenital malformations in the bone injury site.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The population in the surrounding areas of the five centers set up in this study.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The image quality rating scale score. | Immediately after inclusion in the study.
  There are 24 entries in the image quality rating scale with a total score of 100 points. According to the score, there are 4 grades (A. ≥90; B. 80-89; C. 70-79; D. <70), among which D is unqualified.
Difference of fracture detection rate (sensitivity and specificity) between artificial intelligence and expert diagnosis. | Immediately after the diagnosis is completed.
  Sensitivity is the percentage of individuals with bone injury who diagnosed by artificial intelligence or experts. Specificity is the percentage of those without bone injury who have normal diagnosis results.

CONTACTS AND LOCATIONS:
Overall Officials: Guisheng Wang, Doctor, Study Chair — Third center of PLA General Hospital
Locations (4):
- China (4):
  - Center A, Beijing, Beijing Municipality
  - Xucheng He, Neimeng
  - Center C, Xinjiang
  - Center, Xizang

IPD SHARING:
Plan to Share IPD: No